CLINICAL TRIAL: NCT06863636
Title: Efficacy and Safety Study of the Fixed-dose Combination of Celecoxib/Acetaminophen Compared to Celecoxib for the Treatment of Pain in Patients Diagnosed With Osteoarthritis in Acute Exacerbation
Brief Title: Efficacy and Safety of Celecoxib/Acetaminophen Versus Celecoxib for Diagnosed Osteoarthritis in Acute Exacerbation
Acronym: PRECEDENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30221-III-23(1)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Joint Pain; Knee Osteoarthritis; Hip Osteoarthritis
Keywords: Joint pain; Knee Osteoarthritis; Hip Osteoarthritis; Acute pain
MeSH Terms: conditions — Arthralgia; Osteoarthritis, Knee; Osteoarthritis, Hip; Acute Pain | interventions — Celecoxib; Dipeptidyl-Peptidases and Tripeptidyl-Peptidases; Acetaminophen; CelE protein, bacteria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Celecoxib+Acetaminophen (Experimental): Administered orally, 1 tablet a day during 6 weeks
  Interventions: Drug: Celecoxib + Acetaminohen
- Celecoxib + Acetaminophen (Experimental): Administered orally, 1 tablet a day during 6 weeks
  Interventions: Drug: Celecoxi + Acetaminophen
- Celecoxib (Active Comparator): Administered orally, 1 capsule a day during 6 weeks
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib + Acetaminohen — One tablet of 200 mg / 200 mg a day
  Other Names: Cele + Ace
  Arms: Celecoxib+Acetaminophen
Drug: Celecoxi + Acetaminophen — One tablet of 200 mg / 500 mg a day
  Other Names: Cele + Ace
  Arms: Celecoxib + Acetaminophen
Drug: Celecoxib — One capsule of 200 mg a day
  Other Names: Cele
  Arms: Celecoxib

SUMMARY:
This is a Phase III, longitudinal, multicenter, randomized, double-blind clinical trial designed to evaluate the efficacy and safety of a fixed-dose combination of celecoxib and acetaminophen compared to celecoxib monotherapy for the treatment of pain associated with acute exacerbations of osteoarthritis.

DETAILED DESCRIPTION:
Researchers will evaluate the efficacy and safety of a fixed-dose combination of celecoxib and acetaminophen compared to celecoxib monotherapy for the treatment of pain in patients with osteoarthritis experiencing an acute exacerbation over a 6-week follow-up period. Adverse events related to the study interventions will be recorded throughout the follow-up phase.

Participants will:

Be randomized into one of three intervention groups (A, B, or C).

Attend five scheduled clinic visits (Day 0, and Weeks 1, 2, 4, and 6 of follow-up).

Be permitted to take 500 mg of naproxen as rescue medication, if needed, with prior authorization from the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agrees to participate in the study and provides written informed consent.
* Prior diagnosis of knee or hip osteoarthritis based on clinical criteria (according to the American College of Rheumatology (ACR) criteria described in Annex 5).
* Pain in the affected joint with exacerbation lasting no more than 3 weeks.
* Patient reports moderate to severe pain intensity (VAS ≥ 40 mm).
* For women of childbearing potential (a woman is considered fertile after menarche and until postmenopause unless permanently sterile), they must agree to use at least ONE of the following contraceptive methods during the study:

Barrier methods: diaphragm, cervical cap, male condom, female condom, spermicide foam, sponge, or film.

Hormonal methods: combined oral contraceptives, injectable contraceptives, subdermal implant, contraceptive patch.

Intrauterine device (IUD): copper or silver IUD, Levonorgestrel intrauterine system (IUS), and/or combinations of the above as deemed acceptable by the physician.

Women are considered not of childbearing potential if they meet at least ONE of the following criteria:

Postmenopausal. Premenopausal woman with at least ONE of the following: hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.

Male subjects must agree to use a male condom as a contraceptive method during the study.

* At the discretion of the Principal Investigator (PI) or treating physician, the subject has an indication for treatment with the investigational product and may derive clinical benefit from it.

Exclusion Criteria:

* Intolerance or allergy to the investigational product or any of its components (as reported in the medical history and patient interview).
* Participation in another clinical study involving an investigational treatment or participation in one within the last two weeks prior to the study start.
* Potential study bias due to employment or relationship with the research center, sponsor, or being part of a vulnerable population.
* Medical conditions affecting prognosis that prevent outpatient management, to be evaluated by the Principal Investigator for subject inclusion relevance.
* History of advanced, severe, progressive, or unstable disease of any kind that may interfere with efficacy and safety assessments or pose a special risk to the patient.
* Medical contraindication to the investigational product.
* History of allergic reaction to NSAIDs (Non-Steroidal Anti-Inflammatory Drugs), Acetaminophen, or known hypersensitivity to any formulation components.
* Significant gastrointestinal disorders, such as gastric ulcers, Crohn's disease, ulcerative colitis, or gastrointestinal bleeding.
* Prior opioid treatment within the last five days, as reported in the medical history.
* History of treatment failure with COX-2 selective inhibitors, as documented in the medical history.
* History of chronic somatic pain unrelated to knee or hip osteoarthritis (e.g., fibromyalgia, metastatic disease, or Paget's disease).
* History of alcohol or drug abuse within the past year.
* Current treatment with NSAIDs, including COX-2 inhibitors, within the last 72 hours before signing informed consent (except for aspirin used for cardioprotective purposes).
* History of arthroscopy, viscosupplementation, or intra-articular steroid use in the last three months.
* Previous surgery on the affected joint within the last six months.
* Major trauma in the affected joint within the last three weeks.
* History of chronic liver failure (Child-Pugh A, B, or C).
* History of acute or severe renal failure (glomerular filtration rate <30 ml/min/1.73 m²), as reported in the medical history.
* Significant coagulation disorders (e.g., Von Willebrand disease, hemophilia, vitamin K deficiency) or current use of anticoagulants.

Oncologic patients (except basal cell carcinoma) or those with severe illnesses that, according to the investigator, have a poor prognosis or a life expectancy of less than one year, including severe mental illness.

* Patients with symptoms suggestive of active COVID-19 infection (e.g., fever, cough, dyspnea) and/or contact within the last 14 days with a suspected or confirmed COVID-19 patient.
* Positive pregnancy test, pregnant women, those currently breastfeeding, or those planning pregnancy during the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proportion of patients in each treatment group who, based on the baseline assessment, achieved a response according to the OMERACT-OARSI criteria at Weeks 1, 2, 4, and 6 of follow-up. | 6 weeks
  OMERACT (Outcome Measures in Rheumatology) and OARSI (Osteoarthritis Research Society International) jointly developed a core outcome set (COS) for clinical trials in hip and knee osteoarthritis. This COS includes four key domains that should be assessed in all trials: pain, physical function, patient global assessment, and- for studies lasting one year or more-joint imaging. In this study, patients will be evaluated by the researcher at follow-up visits occurring at Weeks 1, 2, 4, and 6.
Number of participants Number of participants reporting treatment-related adverse events, as recorded in the patient diary.treatment-related adverse events through the patient's diary record. | 6 weeks
  To describe the frequency, intensity, and causality of adverse events occurring during the clinical trial, stratified by treatment group. Adverse events will be documented by participants in their patient diaries. Each reported event will be monitored and followed up at the discretion of the investigator.

SECONDARY OUTCOMES:
To analyze the mean change in pain scores, as measured by the WOMAC questionnaire, at Weeks 1, 2, 4, and 6 compared to baseline, by treatment group. | 6 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a disease-specific questionnaire designed to assess physical function, pain, and stiffness in individuals with hip or knee osteoarthritis, based on their experiences over the past 48 hours. In this study, patients will be assessed by the investigator at Weeks 1, 2, 4, and 6 of follow-up.
To analyze the mean change in pain intensity, as measured by the Visual Analog Scale (VAS), at Weeks 1, 2, 4, and 6 compared to baseline, stratified by treatment group. | 6 weeks
  The Visual Analog Scale (VAS) for pain is a straight line where one end represents no pain and the other represents the worst pain imaginable. The investigator will administer the VAS at each visit to assess the patient's pain intensity. At the end of the clinical trial, the percentage change in pain scores will be calculated and compared across treatment groups.
Comparison of the proportion of subjects in each treatment group who achieve a reduction of ≥30% in pain intensity, as measured by the Visual Analog Scale (VAS), at Weeks 1, 2, 4, and 6 compared to baseline. | 6 weeks
  The Visual Analog Scale (VAS) for pain is a unidimensional measurement instrument consisting of a straight line anchored by descriptors, with one end indicating "no pain" and the other representing "the worst pain imaginable." The investigator will administer the VAS at each study visit to evaluate changes in pain intensity. The proportion of patients achieving a pain reduction of more than 30% from baseline will be documented and compared among treatment groups at Weeks 1, 2, 4, and 6.
To analyze the difference in SF-36 quality of life questionnaire scores at six weeks after the initiation of the intervention, compared to baseline, by treatment group. | 6 weeks
  The Short Form-36 (SF-36) is a generic health survey comprising 36 items designed to measure self-reported Health-Related Quality of Life (HRQoL). It evaluates multiple domains of physical and mental health and generates summary scores for both physical and mental components. In this study, the SF-36 questionnaire will be administered to each patient at baseline and again at Week 6 of follow-up.

OTHER OUTCOMES:
To report the treatment adherence rate, expressed as a percentage, for each intervention group. | 6 weeks
  Therapeutic adherence will be defined by the principal investigator. Adherence to treatment will be considered adequate if the patient has taken ≥80% of the prescribed doses by the time of the corresponding evaluation.
To describe the proportion of subjects experiencing therapeutic failure during the study, stratified by treatment group. | 6 weeks
  Therapeutic failure will be defined by the principal investigator following a medical evaluation. The definition requires the presence of all the following criteria: (1) a change in pain intensity of less than 10 mm on the Visual Analog Scale (VAS), or an increase in VAS score compared to baseline; (2) adherence to treatment of ≥80%; (3) a dosing regimen of every 12 hours (i.e., subjects with dose escalation) maintained for at least 7 days; and (4) absence of comorbidities that could contribute to increased pain, such as new trauma or falls.
To report the proportion of patients requiring dose escalation during the follow-up period, stratified by treatment group. | 6 weeks
  At each study visit, dose escalation (one tablet or capsule every 12 hours) may be considered for patients in any of the three treatment arms who meet the following criteria:
  A decrease of less than 10 mm, no change, or an increase in pain intensity on the Visual Analog Scale (VAS) compared to the previous visit.
  Treatment adherence of ≥80%.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel E Rucker-Joerg, MD, Principal Investigator — Clinical Research Institute S.C.; Ivonne A Torres-Quiroz, MD, Principal Investigator — Unidad de Medicina Especializada SMA; Adelfia Urenda-Quezada, MD, Principal Investigator — Servicios Avanzados de Investigación Médica Mediadvance, S.C.; Martha V Chavira-Flores, MD, Principal Investigator — Consultorio Médico "Dr. Rodrigo Suárez Otero"; Rodrigo Suarez-Otero, MD, Principal Investigator — IMACEN S.A. de C.V.
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebrahimzadeh MH, Makhmalbaf H, Birjandinejad A, Keshtan FG, Hoseini HA, Mazloumi SM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) in Persian Speaking Patients with Knee Osteoarthritis. Arch Bone Jt Surg. 2014 Mar;2(1):57-62. Epub 2014 Mar 15. PMID 25207315
- [Background] Puljak L, Marin A, Vrdoljak D, Markotic F, Utrobicic A, Tugwell P. Celecoxib for osteoarthritis. Cochrane Database Syst Rev. 2017 May 22;5(5):CD009865. doi: 10.1002/14651858.CD009865.pub2. PMID 28530031
- [Background] Krieckaert CL, van Tubergen A, Gehin JE, Hernandez-Breijo B, Le Meledo G, Balsa A, Bohm P, Cucnik S, Elkayam O, Goll GL, Hooijberg F, Jani M, Kiely PD, McCarthy N, Mulleman D, Navarro-Compan V, Payne K, Perry ME, Plasencia-Rodriguez C, Stones SR, Syversen SW, de Vries A, Ward KM, Wolbink G, Isaacs JD. EULAR points to consider for therapeutic drug monitoring of biopharmaceuticals in inflammatory rheumatic and musculoskeletal diseases. Ann Rheum Dis. 2023 Jan;82(1):65-73. doi: 10.1136/annrheumdis-2022-222155. Epub 2022 May 12. PMID 35551063
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Busse JW, Bartlett SJ, Dougados M, Johnston BC, Guyatt GH, Kirwan JR, Kwoh K, Maxwell LJ, Moore A, Singh JA, Stevens R, Strand V, Suarez-Almazor ME, Tugwell P, Wells GA. Optimal Strategies for Reporting Pain in Clinical Trials and Systematic Reviews: Recommendations from an OMERACT 12 Workshop. J Rheumatol. 2015 Oct;42(10):1962-1970. doi: 10.3899/jrheum.141440. Epub 2015 May 15. PMID 25979719
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163